CLINICAL TRIAL: NCT06101524
Title: Digital Evaluation of Volumetric Changes of Free Gingival Graft and Gingival Unit Graft With Indirect Method
Brief Title: Volumetric Changes in Free Gingival Graft Procedures Taken With Different Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eda Cetin Ozdemir (Other)
Responsible Party: Sponsor-Investigator, Eda Cetin Ozdemir, assistant professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022/01-01
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Ndirectly Measuring the Difference Between the Free Gingival Graft and the Free Gingival Unit Via a Scanner
Keywords: Free gingival greft; Free gingival unit; Scanner

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Gingival greft Group (Experimental): Patients who are found to have keratinized mucosa insufficiency as a result of the examination, undergo free gingival graft to increase the keratinized mucosa. procedures will be done and you will be called for a check-up after 6 months.
  The keratinized tissue volume formed after the procedure will be evaluated.
  Interventions: Procedure: Free gingival unit, free gingival greft
- Gingival Unit Greft Group (Experimental): Patients who are found to have keratinized mucosa insufficiency as a result of the examination, undergo gingival unit graft to increase the keratinized mucosa. procedures will be done and you will be called for a check-up after 6 months.
  The keratinized tissue volume formed after the procedure will be evaluated.
  Interventions: Procedure: Free gingival unit, free gingival greft

INTERVENTIONS:
Procedure: Free gingival unit, free gingival greft — The free gingival graft and the free gingival unit taken from the upper jaw palatal mucosa were sutured to the lower jaw anterior region.

SUMMARY:
The primary aim of this study is to evaluate the clinical results of free gingival graft and gingival unit graft by indirect method.

To evaluate the 6-month results linearly and volumetrically using an intraoral scanner (TRİOS, 3Shape, Copenhagen, Denmark) (using measurements and on a plaster model).

DETAILED DESCRIPTION:
Deficiency of keratinized tissue includes mucogingival problems among different clinical entities. (Silva et al., 2010) There is no consensus on the minimum amount of attached gingiva required to maintain the health of the gums. However, there are many clinical situations that demonstrate the necessity of keratinized tissue. (Cevallos et al., 2020) (Agarwal et al., 2015) For example, if the attached gingiva is thin, it becomes difficult to perform adequate oral hygiene procedures and plaque. Inflammation and attachment loss are observed due to accumulation. (Gümüş and Buduneli, 2014) (Raoofi et al., 2019) Keratinized tissue width expresses the distance between the coronal margin of the gingival sulcus and the mucogingival line. It is considered to be the main factor in the management and protection of tissue health around natural teeth. (Agudio et al., 2019) Gingival recession refers to the apical displacement of the soft tissue margin from the cemento-enamel border. Oral hygiene and plaque with tooth sensitivity, root caries, unaesthetic appearance as well as loss of periodontal attachment causes retention. (Arzouman et al., n.d.) (Chambrone and Tatakis, 2015) In the treatment of gingival recession Many techniques have been described: Subepithelial connective tissue graft, stemmed grafts (coronally, laterally), free gingival graft (FGG), gingival unit graft (GUG). (Cevallos et al., 2020)(Sriwil et al., 2020). Although significant results are observed, there are different success rates between techniques. (Sriwil et al., 2020) FGG is used not only to cover the root surface but also to increase the width of keratinized tissue. It was first proposed by Nabers for this purpose. (Mörmann et al., 1981) Currently, the FGG's incompatible aesthetic and crude. It has many limitations due to its appearance. (Sriwil et al., 2020)

Due to the limitations of the FGG, there was a need for a new perspective on such phenomena. The vascular characteristics of the graft are important in terms of rapid capillary anastomosis with impaired vascularity of the recipient site. (Sriwil et al., 2020) Gingival sulcus, where thin blood vessels form a network and capillaries show numerous anastomoses is the place. (Jenabian et al., 2016) The vascular plexus of the gingiva, in terms of horizontal anastomoses feeding the marginal zone marginal and interdental tissues to benefit from better blood perfusion of the recipient area can be used, thus increasing the chances of survival of the graft. (Sriwil et al., 2020) (Yıldırım, 2015) The supracrestal part of the gingiva, which includes the marginal and papillary tissues, is included in the soft tissue graft taken to nourish the avascular root surface.

Studies have shown that the marginal, attached, and interdental gingival regions have significantly different vascular distributions. (Sriwil et al., 2020)

Due to these advantages of marginal and interdental tissues, the technique defined as Gingival Unit Graft (GUG) containing marginal and interdental papilla has emerged as an alternative approach to FGG. (Yıldırım, 2015) Kuru and Yıldırım, in their randomized controlled study comparing FGG and GUG in terms of keratinized tissue gain and root surface coverage, reported that DÜG gave better clinical results. (Dry oath Yıldırım, 2013)

G Power 3.1 (University Kiel, Germany) program was used to calculate the effect size. Effect size Free Gingival Graft in the study of Sriwil, Fakher (1) and an effect size of 2.12 d cohen was determined to be sufficient for significance. It was found that a total of 20 samples, at least 10 for each study group, was sufficient with a type 1 error of 0.05 and 99% power.

Free Gingival Graft was applied to 10 patients with keratinized mucosa deficiency, and Gingival Unit Graft was applied to 10 patients. Volumetric changes in the gingiva were measured both clinically and by scanner at the beginning and 6th months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are systemically healty,

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Keratinized gingival width | İnitial and postoperative 6 months
  The change in keratinized tissue width after free gingival graft and gingival graft unit operations was evaluated.
Average gingival thickness change (mm) | İnitial and postoperative 6 months
  The change in average gingival thickness change after free gingival graft and gingival graft unit operations was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Çetin Özdemir, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We have other studies using this data

REFERENCES:
- [Background] Agarwal C, Tarun Kumar AB, Mehta DS. Comparative evaluation of free gingival graft and AlloDerm((R)) in enhancing the width of attached gingival: A clinical study. Contemp Clin Dent. 2015 Oct-Dec;6(4):483-8. doi: 10.4103/0976-237X.169838. PMID 26681852
- [Background] Agudio G, Chambrone L, Selvaggi F, Pini-Prato GP. Effect of gingival augmentation procedure (free gingival graft) on reducing the risk of non-carious cervical lesions: A 25- to 30-year follow-up study. J Periodontol. 2019 Nov;90(11):1235-1243. doi: 10.1002/JPER.19-0032. Epub 2019 Jul 19. PMID 31194255
- [Background] Arzouman A, Deas DE, Mills MP, Huynh-Ba G, Prihoda TJ, Mealey BL. Impact of different surgical protocols on dimensional changes of free soft tissue autografts: A randomized controlled trial. J Periodontol. 2021 Jan;92(1):45-53. doi: 10.1002/JPER.20-0033. Epub 2020 Oct 16. PMID 32716061
- [Background] Cabanes-Gumbau G, Pascual-Moscardo A, Penarrocha-Oltra D, Garcia-Mira B, Aizcorbe-Vicente J, Penarrocha-Diago MA. Volumetric variation of peri-implant soft tissues in convergent collar implants and crowns using the biologically oriented preparation technique (BOPT). Med Oral Patol Oral Cir Bucal. 2019 Sep 1;24(5):e643-e651. doi: 10.4317/medoral.22946. PMID 31422410
- [Background] Cairo F, Nieri M, Cincinelli S, Mervelt J, Pagliaro U. The interproximal clinical attachment level to classify gingival recessions and predict root coverage outcomes: an explorative and reliability study. J Clin Periodontol. 2011 Jul;38(7):661-6. doi: 10.1111/j.1600-051X.2011.01732.x. Epub 2011 Apr 20. PMID 21507033
- [Background] Cevallos CAR, de Resende DRB, Damante CA, Sant'Ana ACP, de Rezende MLR, Greghi SLA, Zangrando MSR. Free gingival graft and acellular dermal matrix for gingival augmentation: a 15-year clinical study. Clin Oral Investig. 2020 Mar;24(3):1197-1203. doi: 10.1007/s00784-019-02983-0. Epub 2019 Jul 12. PMID 31300879
- [Background] De Bruyckere T, Cabeza RG, Eghbali A, Younes F, Cleymaet R, Cosyn J. A randomized controlled study comparing guided bone regeneration with connective tissue graft to reestablish buccal convexity at implant sites: A 1-year volumetric analysis. Clin Implant Dent Relat Res. 2020 Aug;22(4):468-476. doi: 10.1111/cid.12934. Epub 2020 Jul 19. PMID 32686234